CLINICAL TRIAL: NCT03476239
Title: An Open-label, Multicenter, Phase 3 Study to Evaluate Efficacy and Safety of the BiTE Antibody Blinatumomab in Chinese Adult Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Efficacy and Safety of the BiTE Antibody Blinatumomab in Chinese Adult Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130316
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Relapsed; Refractory; B-precursor; Acute Lymphoblastic; Leukemia ALL; Blinatumomab; Chinese Adult Subjects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — blinatumomab

STUDY DESIGN:
Intervention Model Description: Evaluate the efficacy and safety of blinatumomab in Chinese subjects with relapsed/refractory B-precursor ALL, The study will consist of a screening period, a treatment period, and a follow-up period.
  Treatment will consist of up to 5 cycles of blinatumomab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Treatment consisted of two induction cycles and up to 3 consolidation cycles of treatment for responders.
  In the first induction cycle, the initial dose of blinatumomab was 9 μg/day for Days 1-7 and then escalated (dose step) to 28 μg/day starting on day 8 (week 2) through day 29 (week 4). This is followed by two weeks without blinatumomab treatment.
  In subsequent cycles (beginning with the second induction cycle and continuing through consolidation, for applicable participants) 28 μg/day was administered for all 4 weeks of continuous treatment, followed by a treatment-free interval of two weeks.
  Interventions: Drug: Blinatumomab; Drug: Dexamthasone

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab will be supplied as single-use glass injection vials as a sterile, preservative-free, white to off-white, lyophilized powder for reconstitution and administration by continuous intravenous infusion (CIVI).
  A single cycle of blinatumomab treatment is 6 weeks in duration, which includes 4 weeks of blinatumomab CIVI followed by a 2 week treatment-free interval. The treatment-free interval may be prolonged by up to 7 days, if deemed necessary by the investigator.
  Other Names: BLINCYTO®; AMG 103; MT103
Drug: Dexamthasone — Premedication with dexamethasone was intended to prevent cytokine release syndrome (CRS) events associated with blinatumomab treatment. Treatment could start pre-study. Dexamethasone 20 mg IV was administered within 3 hours before start of blinatumomab in each treatment cycle, and within 3 hours before dose step increase.

SUMMARY:
This study is being done to evaluate the rate of hematological response (complete remission/complete remission with partial hematological recovery [CR/CRh*]) induced by blinatumomab in Chinese adults with relapsed/refractory B-precursor acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This is an open label, single-arm, multicenter phase 3 study to evaluate efficacy and safety of the BiTE (bispecific T cell engager) antibody blinatumomab in Chinese adults with relapsed/refractory B-precursor ALL. The study will consist of a screening period, a treatment period, and a follow-up period.

Treatment will consist of up to 5 cycles of blinatumomab. Participants who achieve a bone marrow (BM) response (≤ 5% BM blasts) or CR/CRh*/CRi within 2 induction cycles of treatment may continue to receive up to 3 additional consolidation cycles of blinatumomab. Thirty days after end of the last dose of protocol-specified therapy, participants will have a safety follow-up visit.

If subjects are suitable for allogeneic stem cell transplantation (alloHSCT) after treatment with blinatumomab, they may undergo alloHSCT instead of receiving further consolidation cycles with blinatumomab.

Participants will be followed via clinic visit or telephone contact every 3 months after their safety follow-up visit until death has been observed or a maximum of 2 years after start of treatment, whichever occurs first.

A planned interim analysis to assess efficacy and safety of blinatumomab was to be based on the interim analysis set (N = 90). The efficacious benefit assessment based on an O'Brien-Fleming alpha spending function (O'Brien and Fleming, 1979) with the critical boundary 42.2% at the interim analysis and 39.2% at the primary analysis in CR/CRh* rate. If the interim analysis showed statistically efficacious and overall benefit-risk analysis to be promising per the data review team review, then the interim analysis could become the primary analysis of this study. In addition, the study would continue its enrollment until 120 participants had been enrolled and continued their participation in the study to complete protocol-specified procedures.

The data cutoff date of 12 April 2019 allowed for the 90th participant enrolled before 21 February 2019 to have had the opportunity to complete 2 cycles of treatment and the safety follow-up visit (if the participant had discontinued treatment after 2 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Subjects have provided informed consent/assent prior to initiation of any study-specific activities/procedures or subjects legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
* Subjects with Ph-negative B-precursor ALL, with any of the following:
* Primary refractory after induction therapy or who had relapsed within 12 months of first remission or
* Relapsed within 12 months of receiving allogeneic hematopoietic stem cell transplantation (alloHSCT) or
* Relapsed or refractory after first salvage therapy or beyond
* > 5% blasts in bone marrow (by morphology)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* Age ≥ 18 years at the time of informed consent

Exclusion Criteria:

Disease Related

* Subjects with Ph-positive ALL
* Subjects with Burkitt´s Leukemia according to World Health Organization (WHO) classification.
* History or presence of clinically relevant CNS pathology as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, and psychosis
* Active ALL in the central nervous system (CNS) (confirmed by cerebrospinal fluid [CSF] analysis) or testes
* Isolated extramedullary disease
* Current active autoimmune disease or history of autoimmune disease with potential CNS involvement

Other Medical Conditions

* History of malignancy other than ALL within 5 years prior to start of protocol-specified therapy with the exception of:
* Malignancy treated with curative intent and with no known active disease present for 5 years before enrollment and felt to be at low risk for recurrence by the treating physician.
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated cervical carcinoma in situ without evidence of disease.
* Adequately treated breast ductal carcinoma in situ without evidence of disease.
* Prostatic intraepithelial neoplasia without evidence of prostate cancer.
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive)

Medications or Other Treatments

* Autologous HSCT within 6 weeks prior to start of blinatumomab treatment
* AlloHSCT within 3 months prior to start of blinatumomab treatment
* Any active acute Graft-versus-Host Disease (GvHD), grade 2-4 according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment
* Any systemic therapy against active GvHD within 2 weeks prior to start of blinatumomab treatment
* Cancer chemotherapy within 2 weeks prior to start of blinatumomab treatment (intrathecal chemotherapy and dexamethasone are allowed until start of blinatumomab treatment). In addition, any subject whose organ toxicity (excluding hematologic) from prior ALL treatment has not resolved to common terminology criteria for adverse events (CTCAE) ≤ grade 1.
* Radiotherapy within 2 weeks prior to start of blinatumomab treatment
* Immunotherapy (eg, rituximab) within 4 weeks prior to start of blinatumomab treatment
* Currently receiving treatment in another investigational device or drug study, or less than 4 weeks prior to start of blinatumomab treatment.
* Previous treatment with anti-CD19 therapy

General

* Known hypersensitivity to immunoglobulins or to any other component of the IMP formulation
* Pregnant women and women planning to become pregnant should not participate in this study. Subjects who are breast feeding prior to start of blinatumomab treatment may be enrolled if they stop breast feeding with breast milk produced during blinatumomab treatment and for an additional 48 hours after the last dose of blinatumomab.
* Male participants are not required to use birth control during treatment with blinatumomab. However, you should let your female partner know you are in this study.
* Subject likely to not be available to complete all protocol-required study visits or procedures, including follow-up visits, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the Investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Previous treatment with blinatumomab
* Abnormal screening laboratory values as defined below:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase ALT and/or alkaline phosphatase (ALP) ≥ 5 * upper limit of normal (ULN)
* Total bilirubin (TBL) ≥ 1.5 * ULN (unless related to Gilbert´s or Meulengracht disease)
* Creatinine ≥ 1.5 ULN or creatinine clearance < 60 ml/min (calculated)
* Woman of childbearing potential and is not willing to use 2 effective methods of contraception during treatment and for an additional 48 hours after the last dose of blinatumomab. Birth control is not required for postmenopausal women, or women with uterus/or both ovaries/ or both fallopian tubes removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- China (23):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese People Liberation Army General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi an Jiaotong University, Xi'an, Shaanxi
  - West China Hospital, Sichuang University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital Peking Union Medical College, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Peking University International Hosipital, Beijing
  - Anhui Provincial Hospital, Hefei
  - Huashan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Zhou H, Yin Q, Jin J, Liu T, Cai Z, Jiang B, Li D, Sun Z, Li Y, He Y, Ma L, Gao S, Hu J, He A, Du X, Liu D, Zhang X, Ke X, Zhuang J, Han Y, Wang X, Chen Y, Gordon P, Yu D, Zugmaier G, Wang J. Efficacy and safety of blinatumomab in Chinese adults with Ph-negative relapsed/refractory B-cell precursor acute lymphoblastic leukemia: A multicenter open-label single-arm China registrational study. Hematology. 2022 Dec;27(1):917-927. doi: 10.1080/16078454.2022.2111992. PMID 36000952
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 23 centers in China. The study included a treatment period, a safety follow-up (SFU) visit 30 days after last dose and a follow-up period.
Pre-assignment Details: A pre-specified interim analysis was to occur after the first 90 participants had a chance to complete 2 cycles of treatment and safety follow-up; the data cutoff date for this analysis was 12 April 2019. If the pre-specified efficacious benefit criteria were met, the interim analysis would become the primary analysis.
  A final analysis was conducted once all enrolled participants completed the study.
Groups:
- Blinatumomab: Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. Treatment consisted of two induction cycles and up to 3 consolidation cycles of treatment for responders.
  In the first induction cycle, the initial dose of blinatumomab was 9 μg/day for days 1-7 and then escalated (dose step) to 28 μg/day starting on day 8 (week 2) through day 29 (week 4), followed by two weeks without blinatumomab treatment.
  In subsequent cycles (beginning with the second induction cycle and continuing through consolidation, for applicable participants) 28 μg/day was administered for all 4 weeks of continuous treatment, followed by a treatment-free interval of two weeks.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 121
Received Blinatumomab | 120
Interim Analysis Set (Protocol-specified number of dosed subjects with the opportunity for 2 cycles of treatment) | 90
Completed | 23
Not Completed | 98
Not completed — Withdrawal by Subject | 10
Not completed — Death | 80
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Population: Participants enrolled in the study who received at least 1 infusion of blinatumomab.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (15.2)
Age, Customized [Count of Participants; unit: Participants] — Age group
  Participants
    < 35 years | 71
    ≥ 35 to < 55 years | 31
    ≥ 55 years | 18
Age, Customized [Count of Participants; unit: Participants] — Geriatric age group
  Participants
    < 65 years | 115
    ≥ 65 to < 75 years | 5
    ≥ 75 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 120
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Age at Diagnosis [Mean (Standard Deviation); unit: years] | 34.78 (15.1)
Eastern Cooperative Oncology Group (ECOG) Performance Scale [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  Participants
    Status 0 | 43
    Status 1 | 53
    Status 2 | 24
    Status > 2 | 0
Key Entry Criterion [Count of Participants; unit: Participants] — Criteria #1:Primary refractory or first relapse with remission duration of < 12 months.
  Criteria #2: Relapse any time within 12 months of allo-HSCT (if none of the above).
  Criteria #3: Relapsed or refractory after first salvage therapy or beyond (if none of the above).
  Participants
    Criteria #1 | 70
    Criteria #2 | 10
    Criteria #3 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hematological Response of Complete Remission (CR) or Complete Remission With Partial Hematological Recovery (CRh*) During the First 2 Treatment Cycles With Blinatumomab
Description: A CR is defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts (platelets > 100,000/μL, and absolute neutrophil count [ANC] > 1,000/μL).
  CRh* is defined as ≤ 5% blasts in the bone marrow, no evidence of disease and partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl.
  CR/CRh* rate is defined as the percentage of participants who achieve CR/CRh* within 2 cycles of treatment with blinatumomab. Participants without response assessment were accounted for in the denominator when calculating the response rate, ie, these participants were counted as non-responders.
  The interim analysis was to become the primary analysis by meeting pre-specified efficacy and safety criteria based on an O'Brien-Fleming alpha spending function with the critical boundary 42.2%. Results for both the interim and final analysis are reported.
Time Frame: Within 2 cycles of treatment (12 weeks)
Population: All enrolled participants who received any infusion of blinatumomab. The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
percentage of participants
  Interim Analysis: number analyzed (Participants) | 90
  Interim Analysis | 45.6 [35.0 to 56.4]
  Final Analysis | 48.3 [39.1 to 57.6]

2. Secondary Outcome: Percentage of Participants With a Hematological Response of Complete Remission (CR) During the First 2 Treatment Cycles With Blinatumomab
Description: A CR is defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts (platelets > 100,000/μL, and absolute neutrophil count [ANC] > 1,000/μL).
  CR rate is defined as the percentage of participants who achieved CR within 2 cycles of treatment with blinatumomab. Participants without response assessment were accounted for in the denominator when calculating the response rate, ie, these participants were counted as non-responders.
  Results for both the interim and final analysis are reported.
Time Frame: Within 2 cycles of treatment (12 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
percentage of participants
  Interim Analysis: number analyzed (Participants) | 90
  Interim Analysis | 41.1 [30.8 to 52.0]
  Final Analysis | 43.3 [34.3 to 52.7]

3. Secondary Outcome: Percentage of Participants With a CR or CRh* or Complete Remission With Incomplete Hematological Recovery Without CRh* (CRi) (CR/CRh*/CRi) During the First 2 Treatment Cycles With Blinatumomab
Description: CRi is defined as ≤ 5% blasts in the bone marrow, no evidence of disease and incomplete recovery of peripheral blood counts: platelets > 100,000/μl or ANC > 1,000/μl (but not both).
  CR/CRh*/CRi rate is defined as the percentage of participants who achieve CR/CRh*/CRi within 2 cycles of treatment with blinatumomab. Participants without response assessment were accounted for in the denominator when calculating the response rate, ie, these participants were counted as non-responders.
  Results for both the interim and final analysis are reported.
Time Frame: Within 2 cycles of treatment (12 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
percentage of participants
  Interim Analysis: number analyzed (Participants) | 90
  Interim Analysis | 47.8 [37.1 to 58.6]
  Final Analysis | 50.0 [40.7 to 59.3]

4. Secondary Outcome: Pharmacokinetic (PK) Parameter: Concentration of Blinatumomab at Steady State (Css)
Description: Blinatumomab serum concentration was quantified using a validated enzyme- linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 50 pg/mL.
  Blinatumomab serum steady-state concentrations (Css) was summarized as the average of the observed concentrations collected after 24 hours from the start of continuous IV infusion for each dose level. Cycle 1 day 2 values represent Css for the initial dose of blinatumomab (9 µg/day). Values collected from other time points were used to calculate Css of 28 µg/day dose in their respective cycles.
Time Frame: Cycle 1: Days 2, 15, and 29; Cycle 2: Days 2, 15, and 29 (approximately study days 44, 57, and 71)
Population: Pharmacokinetic analysis set consisting of all participants who received blinatumomab and had at least one PK sample collected. The number of participants analyzed for each time point reflects participants with available Css data; data below the lower limit of quantification and from subjects who did not receive the specified doses were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 118
pg/mL
  Cycle 1: 9 μg/day: number analyzed (Participants) | 94
  Cycle 1: 9 μg/day | 103 (41)
  Cycle 1: 28 μg/day: number analyzed (Participants) | 92
  Cycle 1: 28 μg/day | 416 (72)
  Cycle 2: 28 μg/day: number analyzed (Participants) | 56
  Cycle 2: 28 μg/day | 634 (21)

5. Secondary Outcome: Pharmacokinetic (PK) Parameter: Clearance
Description: Systemic clearance (CL) calculated as the average CL value during cycle 1 and cycle 2, where CL = infusion rate (μg/hour) / Css
Time Frame: Cycle 1: Days 2, 15 and 29; Cycle 2: Days 2, 15 and 29 (approximately study days 44, 57 and 71)
Population: Participants in the pharmacokinetic analysis set with available CL data at at least one post-baseline time point; data below the lower limit of quantification and from participants who did not receive the specified doses were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Blinatumomab
Number analyzed (Participants) | 108
L/hour | 2.86 (57)

6. Secondary Outcome: Pharmacokinetic (PK) Parameter: Terminal Half-Life
Description: Terminal half-life (t1/2,z) calculated as t1/2,z = ln(2)/lambda-z, where lambda-z was the first-order rate constant estimated via linear regression of the terminal log-linear decay phase from day 29 post-end of infusion collections.
Time Frame: Cycle 1 Day 29: prior to end of infusion and after the end of infusion at 3 hours and 6 hours
Population: Participants in the pharmacokinetic analysis set with sufficient data on cycle 1 day 29 to calculate half-life. Data below the lower limit of quantification and from participants who did not receive the specified doses were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Blinatumomab
Number analyzed (Participants) | 9
hours | 2.22 (31)

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Volume of Distribution
Description: The volume of distribution (Vz) was calculated as Vz = CL/lambda-z, where lambda-z was the first-order rate constant estimated based on cycle 1 day 29 collections via linear regression of the terminal log-linear decay phase as determined from the noncompartmental analysis and where CL was the CL averaged over multiple cycles. Volume of distribution was estimated for participants who have sufficient evaluable PK data.
Time Frame: Cycle 1: Days 2, 15 and 29; Cycle 2: Days 2, 15, and 29 (approximately study days 44, 57 and 71)
Population: Participants in the pharmacokinetic analysis set with sufficient data to calculate volume of distribution. Data below the lower limit of quantification and from participants who did not receive the specified doses were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Blinatumomab
Number analyzed (Participants) | 9
liters | 7.15 (61)

8. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival (OS)
Description: Overall survival time was calculated from the time of first infusion of blinatumomab until death due to any cause. Participants still alive were censored at the date last known to be alive up until the data cut-off date (interim analysis) or end of study date (final analysis).
  Months are calculated as days from the first treatment to death/censor date, divided by 30.5.
  Results for both the interim and final analysis are reported.
Time Frame: Interim analysis: From first dose of blinatumomab to the data cutoff date of 12 April 2019; maximum time on follow-up for OS was 14.7 months. Final analysis: From first dose of blinatumomab to end of study; maximum time on follow-up for OS was 25.7 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
months
  Interim Analysis: number analyzed (Participants) | 90
  Interim Analysis | 9.2 [6.5 to 11.7]
  Final Analysis | 9.1 [7.2 to 11.7]

9. Secondary Outcome: Kaplan-Meier Estimate for Relapse-Free Survival (RFS)
Description: Relapse-free survival time was calculated from the first onset of CR/CRh* within the first 2 cycles until the documented hematological relapse, extra-medullary disease, or death due to any cause, whichever occurred first. Participants who were still alive and relapse-free were censored at the date of last disease assessment.
  Months were calculated as days from the first onset of CR/CRh* within the 2 cycles until the documented hematological relapse/extra-medullary disease/death/censor date, divided by 30.5.
  Results for both the interim and final analysis are reported.
Time Frame: Interim Analysis: From first onset of CR/CRh* to the data cutoff date of 12 April 2019; maximum time on follow-up for RFS was 12.4 months. Final Analysis: From first onset of CR/CRh* to end of study; maximum time on follow-up for RFS was 18.1 months.
Population: Enrolled participants who received any infusion of blinatumomab who achieved CR/CRh* during the first 2 cycles. The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit and who achieved CR/CRh* during the first 2 cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 58
months
  Interim Analysis: number analyzed (Participants) | 41
  Interim Analysis | 4.3 [3.2 to 9.4]
  Final Analysis | 5.4 [3.9 to 6.1]

10. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Response During the First Two Treatment Cycles
Description: The detection of MRD (the presence of a low number of leukemic cells that are not detectable by light microscopy) after induction therapy and/or consolidation therapy is an independent prognostic factor for poor outcome of ALL. Participants highly responsive to chemotherapy with a MRD-level < 1 × 10^-4 leukemic cells detectable by flow cytometry induced by induction treatment, have a favorable prognosis.
  MRD response is defined as < 1 ×10^-4 leukemic cells detectable as measured by flow cytometry.
  MRD complete response is defined as having no detectable leukemic cells by flow cytometry.
  Results for both the interim and final analysis are reported.
Time Frame: Within 2 cycles of treatment (12 weeks)
Population: Participants who received any infusion of blinatumomab who achieved CR/CRh* within 2 cycles and had evaluable MRD assessment. The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit who achieved CR/CRh* within 2 cycles and had evaluable MRD assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 58
percentage of participants
  Interim Analysis: MRD Response: number analyzed (Participants) | 41
  Interim Analysis: MRD Response | 82.9 [67.9 to 92.8]
  Interim Analysis: MRD Complete Response: number analyzed (Participants) | 41
  Interim Analysis: MRD Complete Response | 2.4 [0.1 to 12.9]
  Final Analysis: MRD Response | 84.5 [72.6 to 92.7]
  Final Analysis: MRD Complete Response | 1.7 [0.0 to 9.2]

11. Secondary Outcome: Percentage of Participants Who Received an Allogenic Hematopoietic Stem Cell Transplant (alloHSCT) After Achieving CR/CRh* During Treatment
Description: Percentage of participants who underwent allogenic HSCT while in remission among those who responded to treatment by achieving CR/CRh* during treatment.
  Results for both the interim and final analysis are reported.
Time Frame: Interim analysis: Up to the data cutoff date of 12 April 2019; maximum time on follow-up was 14.7 months. Final analysis: Up to the end of study; maximum time on follow-up was 25.7 months.
Population: Enrolled participants who received any infusion of blinatumomab who achieved CR/CRh* during treatment. The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit and who achieved CR/CRh* during treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 58
percentage of participants
  Interim Analysis: number analyzed (Participants) | 41
  Interim Analysis | 22.0 [10.6 to 37.6]
  Final Analysis | 27.6 [16.7 to 40.9]

12. Secondary Outcome: 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplant
Description: The 100-day mortality rate after allogeneic HSCT was defined as the percentage of participants having died up to 100 days after allogeneic HSCT estimated using the estimated time to death in percent calculated by Kaplan-Meier methods. Participants still alive alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive.
Time Frame: 100 days after HSCT
Population: Participants who received any infusion of blinatumomab with a CR/CRh* response who underwent alloHSCT while in remission. The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit, achieved CR/CRh* and underwent alloHSCT while in remission.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 15
percentage of participants
  Interim Analysis: number analyzed (Participants) | 9
  Interim Analysis | 0.0 [NA to NA] — Could not be estimated due to the low number of events
  Final Analysis | 6.7 [1.0 to 38.7]

13. Secondary Outcome: Kaplan-Meier Estimates for Time to a ≥ Ten-Point Decrease From Baseline in Global Health Status Quality of Life
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales, and 9 symptom scales/items. The GHS is reported in this outcome.
  For the GHS, scores range from 0 to 100 with a high score indicating better global health status/functioning. A ≥ 10-point decrease from baseline indicates a deterioration in quality of life.
  Months are calculated from start of blinatumomab date to deterioration/censor date, divided by 30.5.
Time Frame: EORTC QLQ C30 was completed on days 1, 8, 15, and 29 during Cycle 1; days 1, 15, and 29 during cycle 2 and each consolidation cycle, and at the SFU visit (30 days after last dose).
Population: Participants who received blinatumomab treatment and had baseline and ≥ 1 postbaseline result for EORTC QLQ-C30 GHS.
  The interim analysis was based on the first 90 participants who had a chance to complete ≥ 2 cycles of blinatumomab and the safety follow-up visit who had a baseline and ≥ 1 postbaseline result for EORTC QLQ-C30 GHS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 110
months
  Interim Analysis: number analyzed (Participants) | 81
  Interim Analysis | 1.6 [1.0 to NA] — Not enough events to estimate the upper limit
  Final Analysis | 3.7 [1.1 to NA] — Not enough events to estimate the upper limit

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: Adverse events (AEs) were evaluated for severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, as follows:
  Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death.
  An AE was considered "serious" if it resulted in death, was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant incapacity or substantial disruption to conduct normal life functions, was a congenital anomaly or birth defect or was a medically important condition.
Time Frame: From day 1 to 30 days after last infusion of blinatumomab; median (min, max) treatment duration was 30.9 (1, 142) days.
Population: All enrolled participants who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
Participants
  Any TEAE | 120
  TEAE Grade ≥ 3 | 115
  Serious AE | 40
  TEAE leading to drug discontinuation | 18
  Serious AE leading to drug discontinuation | 12
  TEAE leading to drug interruption | 31
  Serious AE leading to drug interruption | 13
  Fatal AE | 11

15. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (TEAE)
Description: Adverse events (AEs) were evaluated for severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, as follows:
  Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death.
  The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
  An AE was considered "serious" if it resulted in death, was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant incapacity or substantial disruption to conduct normal life functions, was a congenital anomaly or birth defect or was a medically important condition.
Time Frame: From day 1 to 30 days after last infusion of blinatumomab; median (min, max) treatment duration was 30.9 (1, 142) days.
Population: All enrolled participants who received any infusion of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 120
Participants
  Any Treatment-related TEAE | 118
  Related TEAE Grade ≥ 3 | 99
  Related Serious AE (SAE) | 29
  Related TEAE leading to drug discontinuation | 16
  Related SAE leading to drug discontinuation | 11
  Related TEAE leading to drug interruption | 25
  Related SAE leading to drug interruption | 10
  Related fatal AE | 6

16. Secondary Outcome: Participants With Anti-Blinatumomab Antibody Formation
Description: Anti-blinatumomab binding antibodies were evaluated with a validated blinatumomab anti-drug antibody assay.
Time Frame: Cycle 2, day 29 (after the completion of Cycle 2) and the SFU visit (30 days after last dose of blinatumomab)
Population: Enrolled participants who received any infusion of blinatumomab with available post-baseline antibody results.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 91
Participants
  Binding antibody positive at anytime | 0
  Neutralizing antibody positive at anytime | 0

ADVERSE EVENTS:
Time Frame: Mortality data are reported from enrollment to the end of study, maximum time on study was 26 months. Adverse events are reported from day 1 to 30 days after last infusion of blinatumomab; the median (min, max) treatment duration was 30.9 (1, 142) days.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 81/121
Serious Adverse Events (participants affected / at risk) | 40/120
Other Adverse Events (participants affected / at risk) | 120/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=120)
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Liver injury (Hepatobiliary disorders) | 3
Cytokine release syndrome (Immune system disorders) | 5
Candida infection (Infections and infestations) | 1
Cytomegalovirus urinary tract infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Haemorrhage intracranial (Nervous system disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Fungaemia (Infections and infestations) | 1
Infection (Infections and infestations) | 1
White blood cell count decreased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=120)
Anaemia (Blood and lymphatic system disorders) | 76
Coagulopathy (Blood and lymphatic system disorders) | 13
Leukocytosis (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 38
Lymphocytosis (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 30
Thrombocytopenia (Blood and lymphatic system disorders) | 37
Abdominal distension (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 15
Haemorrhoids (Gastrointestinal disorders) | 6
Mouth ulceration (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 13
Chest pain (General disorders) | 6
Oedema peripheral (General disorders) | 13
Pyrexia (General disorders) | 57
Hepatic function abnormal (Hepatobiliary disorders) | 12
Liver injury (Hepatobiliary disorders) | 14
Cytokine release syndrome (Immune system disorders) | 71
Infection (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 26
Upper respiratory tract infection (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 7
Activated partial thromboplastin time prolonged (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 28
Albumin globulin ratio increased (Investigations) | 6
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 17
Anion gap increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 32
Beta 2 microglobulin increased (Investigations) | 7
Bilirubin conjugated increased (Investigations) | 18
Blast cell count increased (Investigations) | 7
Blood albumin decreased (Investigations) | 22
Blood alkaline phosphatase increased (Investigations) | 18
Blood bilirubin increased (Investigations) | 23
Blood calcium decreased (Investigations) | 13
Blood fibrinogen decreased (Investigations) | 9
Blood fibrinogen increased (Investigations) | 15
Blood glucose increased (Investigations) | 22
Blood immunoglobulin A decreased (Investigations) | 20
Blood immunoglobulin G decreased (Investigations) | 34
Blood immunoglobulin M decreased (Investigations) | 18
Blood lactate dehydrogenase increased (Investigations) | 54
Blood phosphorus increased (Investigations) | 14
Blood potassium decreased (Investigations) | 10
Blood triglycerides increased (Investigations) | 14
Blood urea increased (Investigations) | 9
Blood uric acid increased (Investigations) | 15
C-reactive protein increased (Investigations) | 60
Eosinophil count decreased (Investigations) | 8
Fibrin D dimer increased (Investigations) | 29
Fibrin degradation products increased (Investigations) | 8
Gamma-glutamyltransferase increased (Investigations) | 33
Globulins decreased (Investigations) | 22
Haematocrit decreased (Investigations) | 7
Haemoglobin decreased (Investigations) | 8
Immunoglobulins decreased (Investigations) | 18
Interleukin level increased (Investigations) | 21
International normalised ratio increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 57
Lymphocyte count increased (Investigations) | 15
Lymphocyte percentage decreased (Investigations) | 11
Lymphocyte percentage increased (Investigations) | 6
Monocyte count decreased (Investigations) | 22
Monocyte percentage decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 58
Neutrophil count increased (Investigations) | 19
Neutrophil percentage decreased (Investigations) | 9
Neutrophil percentage increased (Investigations) | 8
Platelet count decreased (Investigations) | 53
Procalcitonin increased (Investigations) | 21
Protein total decreased (Investigations) | 21
Red blood cell count decreased (Investigations) | 13
Reticulocyte count decreased (Investigations) | 7
Reticulocyte count increased (Investigations) | 17
Serum ferritin increased (Investigations) | 14
Total bile acids increased (Investigations) | 11
White blood cell count decreased (Investigations) | 65
White blood cell count increased (Investigations) | 25
Decreased appetite (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 23
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 15
Hyperuricaemia (Metabolism and nutrition disorders) | 24
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22
Hypocalcaemia (Metabolism and nutrition disorders) | 27
Hypoglycaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 62
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 14
Hypoproteinaemia (Metabolism and nutrition disorders) | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 13
Blood disorder (Blood and lymphatic system disorders) | 6
Sinus tachycardia (Cardiac disorders) | 6
Toothache (Gastrointestinal disorders) | 6
Folliculitis (Infections and infestations) | 6
Blood cholesterol increased (Investigations) | 6
Blood phosphorus decreased (Investigations) | 6
Monocyte count increased (Investigations) | 6
Reticulocyte percentage increased (Investigations) | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT03476239/Prot_002.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT03476239/SAP_001.pdf